CLINICAL TRIAL: NCT00711828
Title: A Phase 2 Clinical Trial of Rituximab, Cyclophosphamide, Bortezomib (VELCADE), and Dexamethasone (R-CYBOR-D) in Relapsed Low Grade and Mantle Cell Lymphoma
Brief Title: Rituximab, Cyclophosphamide, Bortezomib, and Dexamethasone in Treating Patients With Relapsed or Refractory Low-Grade Follicular Lymphoma, Waldenstrom Macroglobulinemia, or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0883; NCI-2011-02991 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0883 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Nodal Marginal Zone Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Bortezomib; Rituximab; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (R-CYBOR-D) (Experimental): Patients receive rituximab IV on day 1and cyclophosphamide PO, bortezomib IV, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Rituximab; Drug: Cyclophosphamide; Drug: Dexamethasone; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Bortezomib — Given IV
Biological: Rituximab — Given IV
  Other Names: MOAB IDEC-C2B8
Drug: Cyclophosphamide — Given PO
Drug: Dexamethasone — Given PO
  Other Names: DM
Other: Questionnaire Administration — Complete a quality of life questionnaire (FACT/GOG neurotoxicity questionnaire, version 4.0)
Other: Quality-of-Life Assessment — Complete a quality of life questionnaire (FACT/GOG neurotoxicity questionnaire, version 4.0)
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial is studying how well giving rituximab and cyclophosphamide together with bortezomib and dexamethasone (R-CyBor-D) works in treating patients with relapsed or refractory low-grade follicular lymphoma, Waldenstrom macroglobulinemia, or mantle cell lymphoma. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab and bortezomib together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess tumor response to R-CyBor-D in patients with relapsed follicular (Gr 1 or 2), mantle cell, marginal zone lymphomas, small lymphocytic lymphoma (SLL)/chronic lymphocytic leukemia (CLL) and lymphoplasmacytic (Waldenstrom's macroglobulinemia) lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate overall survival, progression-free survival, duration of response, and time to treatment failure of patients receiving R-CyBor-D.

II. To describe the adverse event profile (using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v 3.0) of R-CyBor-D.

III. To evaluate quality of life for patient reported neurotoxicity using the Gynecologic Oncology Group's Functional Assessment of Cancer Therapy (FACT/GOG) neurotoxicity questionnaire, version 4.0.

OUTLINE:

Patients receive rituximab intravenously (IV) on day 1and cyclophosphamide orally (PO), bortezomib IV, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of relapsed or refractory follicular Grades 1 or 2 lymphoma, mantle cell lymphoma (MCL), small lymphocytic lymphoma/chronic lymphocytic leukemia (SLL/CLL), extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (MALT) type, nodal marginal zone B-cell lymphoma, splenic marginal zone B-cell lymphoma, or lymphoplasmacytic lymphoma (Waldenstrom's macroglobulinemia/WM) by biopsy ≤ 6 months prior to registration

  * NOTE: MCL diagnosis should be confirmed by cyclin D1 staining or fluorescence in situ hybridization (FISH) (t(11;14))
* Measurable disease by computed tomography (CT), positron emission tomography (PET)/CT or magnetic resonance imaging (MRI) scans with lymph nodes ≥2.0 cm in at least one dimension or tumor cells in the blood ≥ 5 x10^9/L

  * NOTE: Lymphoplasmacytic lymphoma (WM) patients without lymphadenopathy must have 1.) >10% lymphocytes, lymphoplasmacytic cells or plasma cells on a bone marrow aspirate/biopsy, and 2.) quantitative IgM ≥ 400mg/dL
* Expected survival > 3 months
* ECOG Performance Status (PS) 0, 1 or 2
* Absolute Neutrophil Count ≥ 1200
* Platelet ≥ 75000
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 x ULN
* Aspartate aminotransferase (AST) ≤ 3 x ULN
* Creatinine ≤ 1.5 x ULN
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of VELCADE (bortezomib), or agree to completely abstain from heterosexual intercourse
* Male subjects, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Willingness to return to Mayo Clinic institution for follow-up
* Negative serum pregnancy test done <7 days prior to registration, for women of childbearing potential only
* Willingness to complete questionnaires by themselves or with assistance

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women -- confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women;
  * Nursing women;
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse event of the prescribed regimen
* Patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Diagnosed or treated for another malignancy ≤ 3 years prior to registration, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy or low-risk prostate cancer after curative therapy

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* Patient has received other investigational drugs ≤ 14 days prior to registration
* Patient has hypersensitivity to bortezomib, boron or mannitol
* Myocardial infarction ≤ 6 months prior to registration or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities

  * NOTE: Prior to study entry, any electrocardiogram (ECG) abnormality at Screening has to be documented by the investigator as not medically relevant
* Previous cancer therapy, hormonal therapy and surgery < 4 weeks prior to registration
* Patient has ≥ Grade 2 peripheral neuropathy
* Radiation therapy within 3 weeks before randomization

  * Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Reeder, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Rituximab 375 mg/m2 IV on day 1> Cyclophosphamide 300 mg/m2 PO on days 1, 8, 15, 22> Bortezomib 1.3 mg/m2 IV on days 1, 8, 15, 22> Dexamethasone 40 mg PO on days 1, 8, 15, 22
Period: Overall Study
Arm/Group | Treatment
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responses (Complete Response or Partial Response)
Description: A response is defined to be a Complete Response (CR) or Partial Response (PR) noted as the objective status on any evaluation (i.e., best response). The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. A confidence interval for the true success proportion will be calculated according to the properties of the binomial distribution.
Time Frame: up to 12 cycles
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment: Rituximab 375 mg/m2 IV on day 1
  > Cyclophosphamide 300 mg/m2 PO on days 1, 8, 15, 22
  > Bortezomib 1.3 mg/m2 IV on days 1, 8, 15, 22
  > Dexamethasone 40 mg PO on days 1, 8, 15, 22
Arm/Group | Treatment
Number analyzed (Participants) | 21
percentage of participants
  Complete Response (CR) | 19.0 [5.5 to 41.9]
  Partial Response (PR) | 42.9 [21.8 to 66.0]

2. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 21
months | 54.8 [24.6 to 54.8]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival time is defined as the time from registration to the earliest date of documentation of disease progression or death, whichever occurs first. Progression is defines as having any new lesion or increase by 50% of previously involved sites from nadir. The distribution of progression-free survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 21
months | 11.6 [3.8 to NA] — The 95% upper confidence limit was not reached.

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest objective status is first noted to be either a CR or PR to the earliest date progression is documented. MR for Waldenstrom lymphoma will not be included as a response. Median duration of response and the confidence interval for the median duration will be computed.
Time Frame: Up to 3 years from registration
Population: Thirteen patients achieved a CR or a PR and are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 13
months | 25.9 [8 to NA] — The 95% upper confidence limit was not reached.

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. If the patient is considered to be a major treatment violation or is taken off study as a non-protocol failure, the patient will be censored on the date they are removed from treatment. The distribution of time to treatment failure will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 21
months | 6.6 [2 to 11.6]

6. Secondary Outcome: Adverse Events
Description: Adverse events were assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 after each cycle of treatment. The maximum grade for each type of adverse event were recorded for each patient, and frequency tables were reviewed to determine patterns. For this endpoint, the number of patients receiving a Grade 3, Grade 4, or Grade 5 as their highest reported grade regardless of attribution are reported. A full list of adverse events are reported in the Adverse Events section of this report.
Time Frame: up to 12 cycles (28 days per cycle) of treatment
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
participants
  Grade 3 | 19
  Grade 4 | 8
  Grade 5 | 0

ADVERSE EVENTS:
Groups:
- Treatment: Dexamethasone 40 mg PO on days 1, 8, 15, 22
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 7/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Encephalomyelitis infection (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 18 (105)
Cardiac pain (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (15)
Gastritis (Gastrointestinal disorders) | 1 (5)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 20 (111)
Fever (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (2)
Leukocyte count decreased (Investigations) | 17 (63)
Lymphocyte count decreased (Investigations) | 1 (4)
Neutrophil count decreased (Investigations) | 12 (33)
Platelet count decreased (Investigations) | 14 (66)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (97)
Taste alteration (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (8)
Anxiety (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (9)
Cystitis (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes